CLINICAL TRIAL: NCT03913910
Title: Treatment of Perianal Fistulas Through Injection of Autologous and Micro-fragmented Adipose Tissue: a Prospective Multicentre Study
Brief Title: Perianal Fistula Treatment With Autologous Adipose Tissue Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Gabriele Naldini, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: AOUPisana_1
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Perianal Fistula
Keywords: Autologous micro-fragmented adipose tissue; Perianal fistula; Lipogems; Mesenchymal Stem Cells

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lipogems: Lipogems injection in the internal orifice, mucosal, submucosal and muscular layer, in the fistula tract and external orifice.
  Interventions: Procedure: Lipogems

INTERVENTIONS:
Procedure: Lipogems — Autologous micro-fragmented adipose tissue is injected in the internal orifice, mucosal, submucosal and muscular layer, then in the fistula tract and external orifice in addition to anal flap.

SUMMARY:
The study aims to evaluate the efficacy of the local injection of autologous micro-fragmented adipose tissue obtained with the Lipogems®system in patients with trans-sphincteric fistulas untreatable with fistulotomy.

DETAILED DESCRIPTION:
STUDY BACKGROUND

Perianal fistulas are diseases that, by their nature, do not tend to heal spontaneously and are very rarely cured with medical treatment. Their healing is usually pursued through surgery, which often needs to be repeated due to the natural tendency of the fistulas to recur. A surgical treatment that is currently able to provide a high chance of healing is fistulotomy which, however, can injure the anal sphincter and may result in degrading scars and possible fecal incontinence. One possible strategy could be the lipofilling, i.e., autologous adipose tissue transplant containing, among the many, pericytes and progenitor cells, including adult mesenchymal stem cells.

STUDY DESIGN

This is a no profit interventional prospective multicenter study without drugs where 100 patients (10 each participant centre) with a diagnosis of trans-sphincteric anal fistula that is not suitable to be laid open will be enrolled.

After the enrolment, medical history and clinical data will be collected and pre-operatory exams will be performed.

METHODS

- Harvesting of the adipose tissue

The lower/lateral abdomen or, eventually, the inner/outer thigh will be chosen as donor site for adipose tissue harvesting under general or spinal anaesthesia. Before the harvesting, the donor site will be injected with 100 cc of Klein Solution (500 cc saline, 1 cc epinephrine 1/1000 IU, and 40 cc lidocaine 2%) using a disposable 17 gauge blunt cannula connected to a 60-cc luer-lock syringe. The fat will be then harvested (50-100 cc) using a 13 gauge blunt cannula connected to a 20-ml VacLok® syringe.

- Processing of the adipose tissue with the Lipogems® device

The harvested fat will be immediately processed in the Lipogems® processing kit (Lipogems International Spa, Milan, Italy). Lipogems® is a disposable device that mechanically reduces the size of the adipose tissue clusters while eliminating oily substances and blood residues with pro-inflammatory properties. The entire process is carried out in one surgical step in complete immersion in physiological solution minimizing any traumatic action on the cells and microarchitecture. The processed micro-fragmented fat will be collected in a 60-cc syringe and positioned to decant the excess of saline solution. At the end, the product will be transferred in several 5-cc syringes to be re-injected in the patient.

- Surgical procedure and micro-fragmented adipose tissue (Lipogems®) injection

The micro-fragmented autologous adipose tissue will be injected with wheals of no more than 1cc in the internal orifice, mucosal, submucosal and muscular layer, then in the fistula tract and external orifice.

- Follow-up visits and outcome measures

All patients will be assessed at 7 days, 1, 3, 6 and 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged over 18 and under 80 years old.
* Diagnosis, confirmed by standard methods (magnetic resonance and/or trans anal ultrasound), of complex fistula (trans-sphincteric unsuitable for treatment lay-open) without any secondary tracts and no active septic processes, performed 2-4 weeks after the first perianal access drainage procedure and fistulectomy, with positioning of a drainage seton.
* Seton placed at least 4-6 weeks previously
* No previous sphincter saving procedures for the anal fistula
* No limitations to a periodic follow-up lasting for a total of 12 months
* Informed consent form signed

Exclusion Criteria:

* Patients with multiple fistulas
* Active septic process
* Patients unable to follow the pathway required by the protocol
* Patients with active Human Immunodeficiency Virus, Hepatitis B Virus or Hepatitis C Virus infections
* Patients with Irritable Bowel Syndrome
* Patients with rectal-vaginal fistulas
* Patients with a history of cancer lasting less than 5 years
* Patients undergoing cortisone and/or immunosuppressive and/or anticoagulant therapy
* Patients with a history rectal or pelvic radiotherapy
* Pregnant women
* Patients with connective tissue diseases and/or coagulation diseases and/or uncompensated diabetes mellitus
* Failure to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of transphincteric anal fistula that is not suitable to be laid open.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing | 12 months
  Closing of the fistula tract (internal and external orifice)

SECONDARY OUTCOMES:
Safety collecting all types of adverse events | 12 months
  All types of adverse events intra-, peri-, or post-operative will be collected
Pain assessed using the Visual Analogue Scale (VAS) for pain | 12 months
  Pain will be assessed using the Visual Analogue Scale for pain (VAS 0-10), where 0 is no pain and 10 is the maximum pain.
Continence | 12 months
  Continence will be assessed with the Wexner Continence Grading Scale. The score takes into account the type and frequency of incontinence and the extent to which it alters the patient's life.
  This scoring system cross-tabulates frequencies and different anal incontinence presentations (Gas/Liquid/Solid/Pad use/Need for lifestyle alterations) and sums the returned score to a total of 0-20 (where 0 = perfect continence and 20 = complete incontinence).
Patient's satisfaction | 12 months
  Patient's satisfaction will be evaluated using a visual analogue scale 0-5, where 0 is no satisfaction and 5 is maximum satisfaction.
Non inferiority compared with the Advancement flap technique | 12 months
  Non-inferiority will be determined comparing healing rate of Lipogems with retrospective data on the advancement flap.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Pisana - Cisanello, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naldini G, Sturiale A, Fabiani B, Giani I, Menconi C. Micro-fragmented adipose tissue injection for the treatment of complex anal fistula: a pilot study accessing safety and feasibility. Tech Coloproctol. 2018 Feb;22(2):107-113. doi: 10.1007/s10151-018-1755-8. Epub 2018 Feb 16. PMID 29453515
- [Background] Tremolada C, Colombo V, Ventura C. Adipose Tissue and Mesenchymal Stem Cells: State of the Art and Lipogems(R) Technology Development. Curr Stem Cell Rep. 2016;2(3):304-312. doi: 10.1007/s40778-016-0053-5. Epub 2016 Jul 13. PMID 27547712
- [Background] Ceserani V, Ferri A, Berenzi A, Benetti A, Ciusani E, Pascucci L, Bazzucchi C, Cocce V, Bonomi A, Pessina A, Ghezzi E, Zeira O, Ceccarelli P, Versari S, Tremolada C, Alessandri G. Angiogenic and anti-inflammatory properties of micro-fragmented fat tissue and its derived mesenchymal stromal cells. Vasc Cell. 2016 Aug 18;8:3. doi: 10.1186/s13221-016-0037-3. eCollection 2016. PMID 27547374
- [Background] Tremolada C, Ricordi C, Caplan AI, Ventura C. Mesenchymal Stem Cells in Lipogems, a Reverse Story: from Clinical Practice to Basic Science. Methods Mol Biol. 2016;1416:109-22. doi: 10.1007/978-1-4939-3584-0_6. PMID 27236668
- [Background] Vezzani B, Shaw I, Lesme H, Yong L, Khan N, Tremolada C, Peault B. Higher Pericyte Content and Secretory Activity of Microfragmented Human Adipose Tissue Compared to Enzymatically Derived Stromal Vascular Fraction. Stem Cells Transl Med. 2018 Dec;7(12):876-886. doi: 10.1002/sctm.18-0051. Epub 2018 Sep 26. PMID 30255987
- [Background] Garcia-Contreras M, Messaggio F, Mendez AJ, Ricordi C. Metabolomic changes in human adipose tissue derived products following non-enzymatic microfacturing. Eur Rev Med Pharmacol Sci. 2018 May;22(10):3249-3260. doi: 10.26355/eurrev_201805_15088. PMID 29863273
- [Background] Cestaro G, De Rosa M, Massa S, Amato B, Gentile M. Intersphincteric anal lipofilling with micro-fragmented fat tissue for the treatment of faecal incontinence: preliminary results of three patients. Wideochir Inne Tech Maloinwazyjne. 2015 Jul;10(2):337-41. doi: 10.5114/wiitm.2014.47435. Epub 2014 Dec 4. PMID 26240640
- [Background] Bianchi F, Maioli M, Leonardi E, Olivi E, Pasquinelli G, Valente S, Mendez AJ, Ricordi C, Raffaini M, Tremolada C, Ventura C. A new nonenzymatic method and device to obtain a fat tissue derivative highly enriched in pericyte-like elements by mild mechanical forces from human lipoaspirates. Cell Transplant. 2013;22(11):2063-77. doi: 10.3727/096368912X657855. Epub 2012 Oct 8. PMID 23051701
- [Background] Paolella F, Manferdini C, Gabusi E, Gambari L, Filardo G, Kon E, Mariani E, Lisignoli G. Effect of microfragmented adipose tissue on osteoarthritic synovial macrophage factors. J Cell Physiol. 2019 Apr;234(4):5044-5055. doi: 10.1002/jcp.27307. Epub 2018 Sep 6. PMID 30187478